CLINICAL TRIAL: NCT06139042
Title: Early-stage Detection of LIver, Biliary TRAct and PancReatic Cancers by Liquid BiopsY in Periphheral Blood: a Prospective Study (LIBRARY Study)
Brief Title: Early-stage Detection of LIver, Biliary TRAct and PancReatic Cancers
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Guangzhou Burning Rock Dx Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-0871
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Liver Cancer; Biliary Tract Cancer; Pancreatic Cancer
MeSH Terms: conditions — Liver Neoplasms; Biliary Tract Neoplasms; Pancreatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- liver, biliary tract, and pancreatic cancers: participants with liver, biliary tract, and pancreatic cancers
  Interventions: Diagnostic Test: Blood drawing
- liver, biliary tract, and pancreatic benign diseases: participants with liver, biliary tract, and pancreatic benign diseases
  Interventions: Diagnostic Test: Blood drawing
- non-liver, biliary tract, and pancreatic diseases: Participants with no known presence of malignancies or benign diseases
  Interventions: Diagnostic Test: Blood drawing

INTERVENTIONS:
Diagnostic Test: Blood drawing — The participants had their blood drawn.

SUMMARY:
LIBRARY is a prospective, multi-center, observational study aimed at detecting early liver, biliary tract, and pancreatic cancers by combining assays of cell-free DNA (cfDNA) methylation, serum protein, and microRNA.

DETAILED DESCRIPTION:
LIBRARY is a prospective, multi-center, observational study aimed at detecting early liver, biliary tract, and pancreatic cancers by combining assays of cell-free DNA (cfDNA) methylation, serum protein, and microRNA. The study will enroll approximately 458 participants diagnosed with liver, biliary tract, and pancreatic cancers, 330 individuals with corresponding benign diseases and 820 healthy participants.

ELIGIBILITY:
Criteria:

Inclusion Criteria for Cancer Arm Participants:

Age 40-75 years at the day of consenting to the study. Able to provide a written informed consent. Pathologically confirmed liver, biliary tract and pancreatic cancers. No prior or ongoing anti-cancer therapy (local or systematic) prior to study blood draw.

Exclusion Criteria for Cancer Arm Participants:

Pregnancy or lactating women. Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant.

Recipients of blood transfusion within 7 days prior to study blood draw. Recipients of any anti-cancer therapy within 30 days prior to study blood draw, due to diseases other than cancers.

With other known malignant tumors or multiple primary tumors.

Inclusion Criteria for Benign Arm Participants:

Age 40-75 years at the day of consenting to the study. Able to provide a written informed consent. Confirmed diagnosis of benign liver, biliary tract and pancreatic diseases. No prior radical treatment of the benign diseases prior to study blood draw.

Exclusion Criteria for Benign Arm Participants:

Pregnancy or lactating women. Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant.

Recipients of blood transfusion within 7 days prior to study blood draw. Recipients of any anti-cancer therapy within 30 days prior to study blood draw, due to diseases other than cancers.

Confirmed diagnosis of malignancies or precancerous lesion. A history of malignant tumors.

Inclusion Criteria for Healthy Arm Participants:

* Able to provide a written informed consent.
* Able to provide sufficient and qualified blood samples for study tests.
* No cancer related symptoms within 30 days prior to study screening.
* Cancer history with curative treatment completed over 3 years without recurrence prior to study enrollment.

Exclusion Criteria for Healthy Arm Participants:

* Insufficient qualified blood sample for study test.
* During pregnancy or lactation.
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant.
* Recipient of blood transfusion within 30 days prior to study blood draw.
* Recipient of anti-infectious therapy within 14 days prior to study blood draw.
* Have received or are undergoing curative cancer treatment within three years prior to study screening.
* With autoimmune or other diseases with severe comorbidities.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our study included participants diagnosed with liver, biliary tract, and pancreatic cancers or benign diseases as well as participants with no known presence of malignancies or benign diseases.
Sampling Method: Non-Probability Sample
Enrollment: 1608 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of the cfDNA methylation model in detection of liver, biliary tract and pancreatic cancers. | 24 months

SECONDARY OUTCOMES:
The sensitivity and specificity of the combined model in detection of different subtypes of cancers. | 24 months
The sensitivity and specificity of the combined model in detection of different stages of liver, biliary tract and pancreatic cancers. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Weilin Wang, Phd, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No